CLINICAL TRIAL: NCT04321265
Title: Outcomes and Prognostic Factors in Coronavirus Disease (COVID-19) in Very Old Intensive Care Patients
Brief Title: Outcomes and Prognostic Factors in COVID-19
Acronym: COVIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: 20-004
Record Dates: First submitted 2020-03-19; First posted 2020-03-25 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: COVID-19; Elderly Patients; Critical Illness; Survival; Old Age
Keywords: COVID-19; Elderly patients
MeSH Terms: conditions — COVID-19; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim is to study the short-term outcome of elderly ICU patients (≥ 70 years) suffering from COVID-19 using a multicenter and multi-national approach. The secondary aim is to investigate the properties of a simple frailty scale in this cohort, and in particular if this is an instrument that can be used for outcome prediction in this group. In addition, various other parameters of potential relevance for older critically ill patients will be studied.

DETAILED DESCRIPTION:
The study started in March 2020 and included until summer 2021 nearly 4000 patients. Several comprehensive analyses were conducted and published. Subsequently, in December 2021 the protocol was slightly changed and recruitment continues in 2022.

Data are collected regarding: Pre-Admission life conditions with Frailty (Clinical Frailty Scale, CFSF.R.A.I.L Score); vaccination status; ICU-Admission (e.g. SOFA), ICU-Treatment, Survival (30 day and 3 months).

Data are collected electronically through an e-CRF and with baseline documentation of the ICU. The database is located in Denmark, at the Department of Epidemiology, University of Aarhus. Each ICU will only have access through the database of their own patients, and patient ID is not registered (Names, birth-date or social security numbers) so it is in that sense anonymous.

The goal is to recruit at up to 400 ICUs that will continuously collect data. The COVIP Study had two different previous recruitment periods. Period 1 (march to May 2020) finished representing the first wave of the pandemic in most countries. The second recruitment period has been defined being from September 1st to December 31st 2020 representing the second wave in most countries. Recruitment in 2021 also continued until the summer without allocating a specific recruitment period. However, the third recruitment period opened January 1st 2022 and is still ongoing.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 70 years
2. ICU-Admission
3. Infection with SARS-CoV-2

Exclusion Criteria:

1. Age <70 years

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: Patient with Infection with SARS-CoV-2
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-03-19 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Survival | up to 30 days

SECONDARY OUTCOMES:
Frailty | pre-admission
  Frailty will be measured by using the Clinical frailty scale (CFS) a global clinical measure of fitness and frailty in elderly people (1=very fit to 9= terminally ill)

CONTACTS AND LOCATIONS:
Locations (7):
- Department of Intensive Care, Aarhus University Hospital, Aarhus, Denmark
- France (3):
  - Hôpitaux de Paris, Hôpital Saint-Antoine, service de réanimation médicale, Paris
  - INSERM, UMR_S 1136, Institut Pierre Louis d'Epidémiologie et de Santé Publique, Paris
  - Sorbonne Universités, UPMC Univ Paris 06, UMR_S 1136, Institut Pierre Louis d'Epidémiologie et de Santé Publique, Paris
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany
- Norway (2):
  - Department of Anaestesia and Intensive Care, Haukeland University Hospital, Bergen
  - Department of Clinical Medecine,University of Bergen, Bergen

REFERENCES:
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Flaatten H, de Lange DW, Artigas A, Bin D, Moreno R, Christensen S, Joynt GM, Bagshaw SM, Sprung CL, Benoit D, Soares M, Guidet B. The status of intensive care medicine research and a future agenda for very old patients in the ICU. Intensive Care Med. 2017 Sep;43(9):1319-1328. doi: 10.1007/s00134-017-4718-z. Epub 2017 Feb 25. PMID 28238055
- [Background] Flaatten H, De Lange DW, Morandi A, Andersen FH, Artigas A, Bertolini G, Boumendil A, Cecconi M, Christensen S, Faraldi L, Fjolner J, Jung C, Marsh B, Moreno R, Oeyen S, Ohman CA, Pinto BB, Soliman IW, Szczeklik W, Valentin A, Watson X, Zaferidis T, Guidet B; VIP1 study group. The impact of frailty on ICU and 30-day mortality and the level of care in very elderly patients (>/= 80 years). Intensive Care Med. 2017 Dec;43(12):1820-1828. doi: 10.1007/s00134-017-4940-8. Epub 2017 Sep 21. PMID 28936626
- [Background] Rockwood K, Stadnyk K, MacKnight C, McDowell I, Hebert R, Hogan DB. A brief clinical instrument to classify frailty in elderly people. Lancet. 1999 Jan 16;353(9148):205-6. doi: 10.1016/S0140-6736(98)04402-X. No abstract available. PMID 9923878
- [Background] Guidet B, de Lange DW, Boumendil A, Leaver S, Watson X, Boulanger C, Szczeklik W, Artigas A, Morandi A, Andersen F, Zafeiridis T, Jung C, Moreno R, Walther S, Oeyen S, Schefold JC, Cecconi M, Marsh B, Joannidis M, Nalapko Y, Elhadi M, Fjolner J, Flaatten H; VIP2 study group. The contribution of frailty, cognition, activity of daily life and comorbidities on outcome in acutely admitted patients over 80 years in European ICUs: the VIP2 study. Intensive Care Med. 2020 Jan;46(1):57-69. doi: 10.1007/s00134-019-05853-1. Epub 2019 Nov 29. PMID 31784798
- [Background] Katz S, Downs TD, Cash HR, Grotz RC. Progress in development of the index of ADL. Gerontologist. 1970 Spring;10(1):20-30. doi: 10.1093/geront/10.1_part_1.20. No abstract available. PMID 5420677
- [Background] Jung C, Wernly B, Muessig JM, Kelm M, Boumendil A, Morandi A, Andersen FH, Artigas A, Bertolini G, Cecconi M, Christensen S, Faraldi L, Fjolner J, Lichtenauer M, Bruno RR, Marsh B, Moreno R, Oeyen S, Ohman CA, Pinto BB, Soliman IW, Szczeklik W, Valentin A, Watson X, Zafeiridis T, De Lange DW, Guidet B, Flaatten H; VIP1 study group. Electronic address: hans.flaatten@uib.no. A comparison of very old patients admitted to intensive care unit after acute versus elective surgery or intervention. J Crit Care. 2019 Aug;52:141-148. doi: 10.1016/j.jcrc.2019.04.020. Epub 2019 May 2. PMID 31055187
- [Derived] Bruno RR, Wernly B, Artigas A, Fuest K, Schaller SJ, Dannenberg L, Kindgen-Milles D, Kelm M, Beil M, Sviri S, Elhadi M, Joannidis M, Oeyen S, Kondili E, Moreno R, Leaver S, Guidet B, De Lange DW, Flaatten H, Szczeklik W, Jung C; COVIP study group and collaborators on behalf of the COVIP study group. Electronic address: covip@med.uni-duesseldorf.de. Contemporary assessment of short- and functional 90-days outcome in old intensive care patients suffering from COVID-19. J Crit Care. 2025 Apr;86:154984. doi: 10.1016/j.jcrc.2024.154984. Epub 2024 Dec 3. PMID 39631193
- [Derived] Mayerhofer T, Klein S, Wernly B, Flaatten H, Guidet B, De Lange DW, Fjolner J, Leaver S, Beil M, Sviri S, Bruno RR, Artigas A, van Heerden PV, Pinto BB, Schefold JC, Moreno R, Cecconi M, Szczeklik W, Jung C, Joannidis M; COVIP study group. Diabetes mellitus is associated with 90-day mortality in old critically ill COVID-19 patients: a multicenter prospective observational cohort study. Infection. 2023 Oct;51(5):1407-1415. doi: 10.1007/s15010-023-02001-2. Epub 2023 Mar 1. PMID 36854893
- [Derived] Mamandipoor B, Bruno RR, Wernly B, Wolff G, Fjolner J, Artigas A, Pinto BB, Schefold JC, Kelm M, Beil M, Sigal S, Leaver S, De Lange DW, Guidet B, Flaatten H, Szczeklik W, Jung C, Osmani V. COVID-19 machine learning model predicts outcomes in older patients from various European countries, between pandemic waves, and in a cohort of Asian, African, and American patients. PLOS Digit Health. 2022 Nov 8;1(11):e0000136. doi: 10.1371/journal.pdig.0000136. eCollection 2022 Nov. PMID 36812571
- [Derived] Baldia PH, Wernly B, Flaatten H, Fjolner J, Artigas A, Pinto BB, Schefold JC, Kelm M, Beil M, Bruno RR, Binnebossel S, Wolff G, Erkens R, Sigal S, van Heerden PV, Szczeklik W, Elhadi M, Joannidis M, Oeyen S, Marsh B, Andersen FH, Moreno R, Leaver S, De Lange DW, Guidet B, Jung C; COVIP study group. The association of prior paracetamol intake with outcome of very old intensive care patients with COVID-19: results from an international prospective multicentre trial. BMC Geriatr. 2022 Dec 27;22(1):1000. doi: 10.1186/s12877-022-03709-w. PMID 36575394
- [Derived] Wolff G, Wernly B, Flaatten H, Fjolner J, Bruno RR, Artigas A, Pinto BB, Schefold JC, Kelm M, Binneboessel S, Baldia P, Beil M, Sivri S, van Heerden PV, Szczeklik W, Elhadi M, Joannidis M, Oeyen S, Flamm M, Zafeiridis T, Marsh B, Andersen FH, Moreno R, Boumendil A, De Lange DW, Guidet B, Leaver S, Jung C; COVIP Study Group. Sex-specific treatment characteristics and 30-day mortality outcomes of critically ill COVID-19 patients over 70 years of age-results from the prospective COVIP study. Can J Anaesth. 2022 Nov;69(11):1390-1398. doi: 10.1007/s12630-022-02304-2. Epub 2022 Aug 9. PMID 35945477
- [Derived] Polok K, Fronczek J, Artigas A, Flaatten H, Guidet B, De Lange DW, Fjolner J, Leaver S, Beil M, Sviri S, Bruno RR, Wernly B, Bollen Pinto B, Schefold JC, Studzinska D, Joannidis M, Oeyen S, Marsh B, Andersen FH, Moreno R, Cecconi M, Jung C, Szczeklik W; COVIP Study Group. Noninvasive ventilation in COVID-19 patients aged >/= 70 years-a prospective multicentre cohort study. Crit Care. 2022 Jul 22;26(1):224. doi: 10.1186/s13054-022-04082-1. PMID 35869557
- [Derived] Bruno RR, Wernly B, Flaatten H, Fjolner J, Artigas A, Baldia PH, Binneboessel S, Bollen Pinto B, Schefold JC, Wolff G, Kelm M, Beil M, Sviri S, van Heerden PV, Szczeklik W, Elhadi M, Joannidis M, Oeyen S, Kondili E, Marsh B, Wollborn J, Andersen FH, Moreno R, Leaver S, Boumendil A, De Lange DW, Guidet B, Jung C; COVIP study group. The association of the Activities of Daily Living and the outcome of old intensive care patients suffering from COVID-19. Ann Intensive Care. 2022 Mar 18;12(1):26. doi: 10.1186/s13613-022-00996-9. PMID 35303201
- [Derived] Bruno RR, Wernly B, Wolff G, Fjolner J, Artigas A, Bollen Pinto B, Schefold JC, Kindgen-Milles D, Baldia PH, Kelm M, Beil M, Sviri S, van Heerden PV, Szczeklik W, Topeli A, Elhadi M, Joannidis M, Oeyen S, Kondili E, Marsh B, Andersen FH, Moreno R, Leaver S, Boumendil A, De Lange DW, Guidet B, Flaatten H, Jung C; COVIP study group. Association of chronic heart failure with mortality in old intensive care patients suffering from Covid-19. ESC Heart Fail. 2022 Jun;9(3):1756-1765. doi: 10.1002/ehf2.13854. Epub 2022 Mar 10. PMID 35274490
- [Derived] Guidet B, Jung C, Flaatten H, Fjolner J, Artigas A, Pinto BB, Schefold JC, Beil M, Sigal S, van Heerden PV, Szczeklik W, Joannidis M, Oeyen S, Kondili E, Marsh B, Andersen FH, Moreno R, Cecconi M, Leaver S, De Lange DW, Boumendil A; VIP2 and COVIP study groups. Increased 30-day mortality in very old ICU patients with COVID-19 compared to patients with respiratory failure without COVID-19. Intensive Care Med. 2022 Apr;48(4):435-447. doi: 10.1007/s00134-022-06642-z. Epub 2022 Feb 26. PMID 35218366
- [Derived] Jung C, Mamandipoor B, Fjolner J, Bruno RR, Wernly B, Artigas A, Bollen Pinto B, Schefold JC, Wolff G, Kelm M, Beil M, Sviri S, van Heerden PV, Szczeklik W, Czuczwar M, Elhadi M, Joannidis M, Oeyen S, Zafeiridis T, Marsh B, Andersen FH, Moreno R, Cecconi M, Leaver S, De Lange DW, Guidet B, Flaatten H, Osmani V. Disease-Course Adapting Machine Learning Prognostication Models in Elderly Patients Critically Ill With COVID-19: Multicenter Cohort Study With External Validation. JMIR Med Inform. 2022 Mar 31;10(3):e32949. doi: 10.2196/32949. PMID 35099394
- [Derived] Polok K, Fronczek J, van Heerden PV, Flaatten H, Guidet B, De Lange DW, Fjolner J, Leaver S, Beil M, Sviri S, Bruno RR, Wernly B, Artigas A, Pinto BB, Schefold JC, Studzinska D, Joannidis M, Oeyen S, Marsh B, Andersen FH, Moreno R, Cecconi M, Jung C, Szczeklik W; COVIP study group. Association between tracheostomy timing and outcomes for older critically ill COVID-19 patients: prospective observational study in European intensive care units. Br J Anaesth. 2022 Mar;128(3):482-490. doi: 10.1016/j.bja.2021.11.027. Epub 2021 Nov 29. PMID 34955167
- [Derived] Jung C, Flaatten H, de Lange D, Beil M, Guidet B. The relationship between treatment limitations and pressure on intensive care units in elderly patients. Intensive Care Med. 2022 Jan;48(1):124-125. doi: 10.1007/s00134-021-06553-5. Epub 2021 Nov 5. No abstract available. PMID 34741189
- [Derived] Jung C, Fjolner J, Bruno RR, Wernly B, Artigas A, Bollen Pinto B, Schefold JC, Wolff G, Kelm M, Beil M, Sviri S, van Heerden PV, Szczeklik W, Czuczwar M, Joannidis M, Oeyen S, Zafeiridis T, Andersen FH, Moreno R, Leaver S, Boumendil A, De Lange DW, Guidet B, Flaatten H; , COVIP Study Group. Differences in mortality in critically ill elderly patients during the second COVID-19 surge in Europe. Crit Care. 2021 Sep 23;25(1):344. doi: 10.1186/s13054-021-03739-7. PMID 34556171
- [Derived] Bruno RR, Wernly B, Flaatten H, Fjolner J, Artigas A, Bollen Pinto B, Schefold JC, Binnebossel S, Baldia PH, Kelm M, Beil M, Sigal S, van Heerden PV, Szczeklik W, Elhadi M, Joannidis M, Oeyen S, Zafeiridis T, Wollborn J, Arche Banzo MJ, Fuest K, Marsh B, Andersen FH, Moreno R, Leaver S, Boumendil A, De Lange DW, Guidet B, Jung C; COVIP Study Group. Lactate is associated with mortality in very old intensive care patients suffering from COVID-19: results from an international observational study of 2860 patients. Ann Intensive Care. 2021 Aug 21;11(1):128. doi: 10.1186/s13613-021-00911-8. PMID 34417919
- [Derived] Jung C, Flaatten H, Fjolner J, Bruno RR, Wernly B, Artigas A, Bollen Pinto B, Schefold JC, Wolff G, Kelm M, Beil M, Sviri S, van Heerden PV, Szczeklik W, Czuczwar M, Elhadi M, Joannidis M, Oeyen S, Zafeiridis T, Marsh B, Andersen FH, Moreno R, Cecconi M, Leaver S, Boumendil A, De Lange DW, Guidet B; COVIP study group. The impact of frailty on survival in elderly intensive care patients with COVID-19: the COVIP study. Crit Care. 2021 Apr 19;25(1):149. doi: 10.1186/s13054-021-03551-3. PMID 33874987
- [Derived] Jung C, Bruno RR, Wernly B, Joannidis M, Oeyen S, Zafeiridis T, Marsh B, Andersen FH, Moreno R, Fernandes AM, Artigas A, Pinto BB, Schefold J, Wolff G, Kelm M, De Lange DW, Guidet B, Flaatten H, Fjolner J; COVIP study group. Inhibitors of the renin-angiotensin-aldosterone system and COVID-19 in critically ill elderly patients. Eur Heart J Cardiovasc Pharmacother. 2021 Jan 16;7(1):76-77. doi: 10.1093/ehjcvp/pvaa083. No abstract available. PMID 32645153
- See also: Related Info — http://vipstudy.org/covip-study/